CLINICAL TRIAL: NCT04459130
Title: Effectiveness of School-Based Weight Management Program in Overweight and Obese Children Between 8-11 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, nesrin arslan, lecturer, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-196
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Childhood Obesity; Child Obesity
Keywords: childhood obesity; school based; obesity intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Child Obesity Program (COP), The program consists of 10 sessions, each lasting 40 minutes. An EOP booklet containing session programs will be distributed to children.The research was determined as randomized controlled pretest-posttest control group design type.
Who Masked: Participant
Masking Description: participants do not know they are in the experimental or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Obesity Program (Experimental): Firstly, overweight and obese students will be determined by measuring their height and weight. While selecting children for the experimental group, random numbers table will be used. As a result of statistical analysis, 33 students will be selected to the Experiment group. Child Obesity Program (COP) will be applied to students in the experimental group for 10 weeks. Before the program is implemented, children's height, weight, subcutaneous adipose tissue measurements will be made. The pedometer wristband will be distributed.
  Pretest: BMI, weight average, subcutaneous adipose tissue measurement and application of scales
  * - Children's Dietary Self- Efficacy Scale-CDSS
  * - Food Behavior Scale
  * - Child Heart Health Development Attitude Scale (exercise, stress, nutrition subscales)
  * -Daily Food Consumption Form
  * -Drink Consumption Form
  * Health Perception Form
  Follow-ups will be performed in the 6th and 9th months after the intervention
  Interventions: Behavioral: Child Obesity Program
- Control Grup (No Intervention): Firstly, overweight and obese students will be determined by measuring their height and weight. When selecting children for the control group, random numbers table will be used. As a result of statistical analysis, 33 students will be selected to the Control group. First, children's height, weight, subcutaneous adipose tissue measurements will be made. The pedometer wristband will be distributed. The control group will be trained for a daily healthy diet and physical activity.
  Pretest: BMI, weight average, subcutaneous adipose tissue measurement and application of scales
  * - Children's Dietary Self- Efficacy Scale-CDSS
  * - Food Behavior Scale
  * - Child Heart Health Development Attitude Scale (exercise, stress, nutrition subscales)
  * -Daily Food Consumption Form
  * -Drink Consumption Form
  * Health Perception Form
  Follow-ups will be performed in the 6th and 9th months after the intervention

INTERVENTIONS:
Behavioral: Child Obesity Program — The program consists of 10 sessions, each lasting 40 minutes. An EOP booklet containing session programs will be distributed to children.
  The topics of the sessions are as follows:
  Session 1: Healthy lifestyles
  * Session 2: Self-esteem and positive thinking, Setting goals Session 3: Stress and Coping, Coping with Emotions in Healthy Ways Session 4: Personality and effective communication
  * Session 5: Activity: Time for action Session 6: Nutrition basics Session 7: Reading tags Session 8: Portion size, nutrition and healthy food choices in schools Session 9: Snacks can also be healthy: Healthy choices
  * Session 10: Together for a healthy life (Melnyk et al., 2006; 2007; 2009). Detailed information about the sessions is given in annex -3.
  Arms: Child Obesity Program

SUMMARY:
Obesity, which is an important public health problem of the last century globally, affects not only adults but also children and young people. Reducing childhood obesity requires effective lifestyle changes and behavioral interventions aimed at healthy nutrition, physical activity and stress management.

to reduce childhood obesity, including school-based multi-component behavioral research in Turkey it has not been demonstrated to parents.

The program, which is planned to be carried out and aims to reduce overweight and obesity in children, is a school-based parenting lifestyle intervention involving multiple behaviors. The program includes family visits, game-based physical activity activities with children, healthy eating recommendations and healthy eating activities with parent participation. The program planned to be implemented was developed to evaluate whether healthy preferences and lifestyle intervention reduce obesity. The aim of this study is to make the positive health behaviors permanent in children, to be a guide for combating childhood obesity and to be useful for future research. to be applied to the research, nutrition consists of 10 sessions, physical activity, including issues such as coping with healthy ways with stress Child Obesity Program (COP), it is thought to overcome this deficiency was needed in Turkey.

ELIGIBILITY:
Inclusion Criteria:

- Overweight or obese children aged 8-11

* Volunteers to participate in the research
* Students who are allowed to participate in the research by their parents

Exclusion Criteria:

* Children with any physical or mental disability and chronic disease (diabetes, metabolic syndrome, heart disease… etc)

  * Children who have normal weight
  * Children who constantly use the drug that can affect weight management (weight gain and loss) The age group included in the study Piaget's development theory coincides with the concrete process period. Concrete

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
BKI, | through study completion, an average of 1 year
  Up to 1 year BKI reduction expected at the end of the program
Subcutaneous adipose tissue | through study completion, an average of 1 year
  Up to 1 year BKI reduction expected at the end of the program

SECONDARY OUTCOMES:
number of steps | through study completion, an average of 1 year
  An increase is expected at the end of the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No